CLINICAL TRIAL: NCT00880126
Title: Community Development Teams to Scale-Up MTFC in California
Brief Title: Community Development Teams to Scale-Up Multidimensional Treatment Foster Care (MTFC) in California
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Center for Research to Practice (Other)
Responsible Party: Patricia Chamberlain, Ph.D., Center for Research to Practice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH076158 (NIH)
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2009-04-13 (Estimated); Status verified 2009-02

CONDITIONS: Behavior Problems
Keywords: Individualized Implementation; Community Development Teams
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CDT (Experimental): Community Development Teams bring together counties who are implementing a new practice
  Interventions: Behavioral: Community Development Teams

INTERVENTIONS:
Behavioral: Community Development Teams — CDTs bring together counties who are implementing a new practice

SUMMARY:
The effects of using Community Development Teams to increase the number of counties that successfully implement and sustain Multidimensional Treatment Foster Care programs is studied in a randomized trial in 40 California counties. MTFC is an alternative to group or residential placement for youth with severe conduct and emotional problems referred from the juvenile justice and child welfare systems.

ELIGIBILITY:
Inclusion Criteria:

* Non-early adopters of evidence-based practice (MTFC)

Exclusion Criteria:

* Placed fewer than 6 youth per year in group care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2006-09; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Implementation of an evidence-based practice in counties | 5 years

REFERENCES:
- [Derived] Brown CH, Chamberlain P, Saldana L, Padgett C, Wang W, Cruden G. Evaluation of two implementation strategies in 51 child county public service systems in two states: results of a cluster randomized head-to-head implementation trial. Implement Sci. 2014 Oct 14;9:134. doi: 10.1186/s13012-014-0134-8. PMID 25312005
- [Derived] Palinkas LA, Holloway IW, Rice E, Brown CH, Valente TW, Chamberlain P. Influence network linkages across implementation strategy conditions in a randomized controlled trial of two strategies for scaling up evidence-based practices in public youth-serving systems. Implement Sci. 2013 Nov 14;8:133. doi: 10.1186/1748-5908-8-133. PMID 24229373
- [Derived] Palinkas LA, Holloway IW, Rice E, Fuentes D, Wu Q, Chamberlain P. Social networks and implementation of evidence-based practices in public youth-serving systems: a mixed-methods study. Implement Sci. 2011 Sep 29;6:113. doi: 10.1186/1748-5908-6-113. PMID 21958674